CLINICAL TRIAL: NCT03340064
Title: An Open-Label, Single-Arm, Multicenter Study of Levetiracetam as Monotherapy or Adjunctive Treatment of Partial Seizures in Pediatric Epileptic Subjects Ranging From 1 Month to Less Than 4 Years of Age
Brief Title: A Study of Levetiracetam as Monotherapy or Adjunctive Treatment of Partial Seizures in Pediatric Epileptic Subjects Ranging From 1 Month to Less Than 4 Years of Age
Acronym: PEACH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Japan Co. Ltd. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EP0100
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Results first posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Partial Seizures
Keywords: Epilepsy; Partial Seizures; Levetiracetam; Monotherapy; Adjunctive Treatment
MeSH Terms: conditions — Seizures; Epilepsy | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Levetiracetam (Experimental): Subjects aged 1 month to <6 months will be started on levetiracetam (LEV) 14 mg/kg/day at Visit 3. The dose may be increased by LEV 14 mg/kg/day for subjects aged 1 month to <6 months at 2-week intervals to a maximum dose of 42 mg/kg/day. Subjects aged 6 months to <4 years will be started on LEV 20 mg/kg/day at Visit 3. The dose may be increased by LEV 20 mg/kg/day at 2-week intervals to a maximum dose of 60 mg/kg/day.
  At Visit 6, subjects may enter the Second Period or enter the Down-Titration Period followed by a Safety Follow-Up Period. Subjects who do not enter the Second Period will be down-titrated. The dose will be decreased by LEV 14 mg/kg/day for subjects aged 1 month to <6 months or by LEV 20 mg/kg/day for subjects aged 6 months to <4 years at 2-week intervals to 0 mg/kg/day.
  Interventions: Drug: Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam — levetiracetam dry syrup 50% for oral administration and levetiracetam solution for infusion (100 mg/mL)
  Other Names: Keppra; E-Keppra; LEV

SUMMARY:
This is a study to confirm the efficacy of levetiracetam as adjunctive treatment or as monotherapy in pediatric epilepsy subjects aged 1 month to less than 4 years of age with partial seizures.

DETAILED DESCRIPTION:
The study will consist of 2 periods. The First Period (6 weeks drug treatment) is designed to confirm efficacy of levetiracetam (LEV), and the Second Period is designed to evaluate the long-term efficacy and safety of LEV.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have a diagnosis of epilepsy with partial onset seizures whether or not secondarily generalized
* Male or female from 1 month to <4 years of age. Pre-term infants aged <1 year are to be stratified into an appropriate age category using the best estimate of their corrected gestational age
* For subjects on adjunctive therapy, subject must be on a stable antiepileptic drug (AED) regimen for the Selection and Evaluation Periods of the study. Minor adjustments to the dose of current AEDs are allowed only prior to Visit 1. Monotherapy subjects must not receive AED treatment, receive temporary AED treatment, or switch an AED prior to Visit 1
* Subject weighs >=3.0 kg
* Subject may have Vagal Nerve Stimulation (VNS) which has been implanted for at least 6 months prior to Visit 1; the settings must be stable for at least 2 months prior to Visit 1. Activated VNS must be counted as 1 of the 2 AEDs
* Subject must have experienced at least 2 observable partial seizures, with or without secondary generalization during each 7-day period during the 2 weeks prior to Visit 1. This time period (the 2 weeks prior to Visit 1) will be referred to as the Retrospective Baseline Period. This seizure information (including type, frequency, and date) must have been recorded on a daily record card (DRC) in order to be acceptable
* If epilepsy surgery has been performed prior to study entry, subjects must have a documented failed epilepsy surgery outcome at least 4 weeks prior to Visit 1
* The use of intermittent benzodiazepines, phenobarbitals, and phenytoins is allowed as long as the frequency is not greater than 1 single administration per week for at least 2 weeks prior to Visit 1 and throughout study participation. If benzodiazepines are used more than once a week, they must be considered as 1 of the AEDs

Exclusion Criteria:

* Subject has been taking any medication (other than their concomitant AEDs) that influences the central nervous system (CNS) for which they had not been on a stable regimen for at least 1 month prior to Visit 1
* Subject is taking any medication that may interfere with the absorption, distribution, metabolism, or excretion of the concomitant AEDs or levetiracetam (LEV) during the course of the study
* Subject has received any investigational medication or device within 30 days prior to Visit 1
* Subject has taken LEV prior to the study
* Subjects using felbamate who have presented with clinically significant abnormalities and/or hepatic function during felbamate treatment, and subjects who are taking felbamate <1year from the date of Visit 1
* History of status epilepticus requiring hospitalization during the 30 days prior to Visit 1, except for status epilepticus occurring during the first 10 days of life
* Subject has a treatable seizure etiology
* Subject is on a ketogenic diet (concomitantly or within 30 days prior to Visit 1)
* Subject has epilepsy secondary to progressing cerebral diseases
* Subject has a current diagnosis of Rasmussen's syndrome, Landau-Kleffner disease or Lennox-Gastaut syndrome
* Clinically significant deviations from reference range values for renal function or any of the other laboratory parameters required for this study, as determined by the Investigator
* Clinically significant acute or chronic illness (as determined during the physical examination or from other information available to the Investigator)
* Allergy to pyrrolidine derivatives or a history of multiple drug allergies
* Subject is known to have a terminal illness
* Subject has a disorder or condition that may interfere with the absorption, distribution, metabolism, or excretion of medications
* Subject has a history of or presence of pseudoseizures
* Subject has any medical condition that might interfere with the subject's study participation
* Subject has ≥3x upper limit of normal (ULN) of any of the following: alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), or >ULN total bilirubin (≥1.5xULN total bilirubin if known Gilbert's syndrome). If subject has elevations only in total bilirubin that are >ULN and <1.5xULN, fractionate bilirubin to identify possible undiagnosed Gilbert's syndrome (ie, direct bilirubin <35%)

Ages: 1 Month to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2023-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (21):
- Japan (21):
  - Ep0100 15, Fukuoka
  - EP0100 3, Hamamatsu
  - EP0100 6, Izumi
  - Ep0100 20, Kobe
  - EP0100 2, Kodaira
  - Ep0100 21, Kofu
  - EP0100 7, Kōshi
  - EP0100 9, Nagakute
  - EP0100 5, Niigata
  - Ep0100 14, Okayama
  - Ep0100 13, Osaka
  - Ep0100 12, Ōbu
  - Ep0100 11, Ōmura
  - Ep0100 18, Saitama
  - EP0100 4, Sapporo
  - Ep0100 10, Sendai
  - Ep0100 19, Sendai
  - Ep0100 16, Shinjuku-ku
  - Ep0100 17, Shinjuku-ku
  - EP0100 1, Shizuoka
  - Ep0100 22, Toyoake

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed.All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://www.Vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in November 2017 and concluded in July 2023.
Pre-assignment Details: Participant Flow refers to the Safety Set Adjunctive therapy (SS_A) and Safety Set Monotherapy (SS_M).
Groups:
- Levetiracetam: Adjunctive Therapy: Participants aged 1 month to less than (<) 6 months received Levetiracetam (LEV) 14 milligram per kilogram per day (mg/kg/day) as adjunctive therapy at Visit 3 (Week 0) of First Period and dose up titrated up to 42 mg/kg/day. Participants aged 6 months to <4 years received LEV 20 mg/kg/day at Visit 3 (Week 0) of first period and dose up titrated up to a maximum of 60 mg/kg/day up to 6 weeks. The dose was increased by 2 weeks interval as per Investigator's discretion. At Visit 6 (Week 6), dose of participants either down-titrated during 4 weeks interval or they entered in second period and continued LEV 14 to 42 mg/kg/day in participants aged 1 month to <6 months or LEV 20 to 60 mg/kg/day for participants aged greater than or equal to (≥) 6 months <4 years at the discretion of the Investigator. Participants visited every 4 weeks for the first 6 months of administration and then every 12 weeks thereafter until approval or till program discontinued. The dose down-titrated during 4 weeks Interval at the discretion of Investigator.
- Levetiracetam: Monotherapy: Participants aged 1 month to < 6 months received LEV 14 mg/kg/day as monotherapy at Visit 3 (Week 0) of First Period and dose up titrated up to 42 mg/kg/day. Participants aged 6 months to <4 years received LEV 20 mg/kg/day at Visit 3 (Week 0) of first period and dose up titrated up to a maximum of 60 mg/kg/day up to 6 weeks. The dose was increased by 2 weeks interval as per Investigator's discretion. At Visit 6 (Week 6), dose of participants either down-titrated during 4 weeks interval or they entered in second period and continued LEV 14 to 42 mg/kg/day in participants aged 1 month to <6 months or LEV 20 to 60 mg/kg/day for participants aged ≥ 6 months <4 years at the discretion of the Investigator. Participants visited every 4 weeks for the first 6 months of administration and then every 12 weeks thereafter until approval or till the program discontinued. The dose could be down-titrated during 4 weeks Interval at the discretion of Investigator.
Period: First Period
Arm/Group | Levetiracetam: Adjunctive Therapy | Levetiracetam: Monotherapy
Started | 32 | 6
Completed | 27 | 6
Not Completed | 5 | 0
Not completed — Adverse Event, non-fatal | 2 | 0
Not completed — Lack of Efficacy | 3 | 0
Period: Second Period
Arm/Group | Levetiracetam: Adjunctive Therapy | Levetiracetam: Monotherapy
Started | 27 | 6
Completed | 8 | 4
Not Completed | 19 | 2
Not completed — Adverse Event, non-fatal | 1 | 1
Not completed — Lack of Efficacy | 11 | 0
Not completed — Physician Decision | 3 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Approved Drug Available For Indication | 1 | 0
Not completed — Protocol-Specified Withdrawal Criterion Met | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the SS_A and SS_M. The SS_A consisted of all enrolled participants on adjunctive therapy who received at least 1 dose of study medication in the evaluation period. The SS_M consisted of all enrolled participants on monotherapy who received at least 1 dose of study medication in the evaluation period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Levetiracetam: Adjunctive Therapy | Levetiracetam: Monotherapy | Total
Number analyzed (Participants) | 32 | 6 | 38
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.7 (10.7) | 32.4 (13.2) | 17.5 (12.7)
Age, Customized [Count of Participants; unit: Participants]
  28 days - <24 months | 26 | 3 | 29
  24 months - <12 years | 6 | 3 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 5 | 20
  Male | 17 | 1 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 32 | 6 | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japan | 32 | 6 | 38

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Partial Seizure Frequency Per Week From Baseline to Visit 6
Description: The percent difference in partial seizure frequency per week at Baseline and Study Visit 6 (Week 6) was computed as: {[(Number of partial seizures per week at Baseline) minus (Number of partial seizures per week at Study Visit 6)] divided by (Number of partial seizures per week at Baseline)} multiplied by 100. A positive value in percent difference from Baseline indicates a reduction in partial seizure frequency from Baseline. Data of this outcome measure was analyzed and reported for participants on adjunctive therapy.
Time Frame: From Baseline (Week 0) to Visit 6 (up to Week 6)
Population: The Full Analysis Set Adjunctive therapy (FAS_A) consisted of all participants in the SS_A who had at least 1 post-Baseline efficacy assessment. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: percent change
Arm/Group | Levetiracetam: Adjunctive Therapy
Number analyzed (Participants) | 28
percent change | 24.24 [-25.48 to 51.85]

2. Secondary Outcome: Percent Change in Partial Seizure Frequency Per Week From Baseline to Visit 4
Description: The percent difference in partial seizure frequency per week at Baseline and Study Visit 4 (Week 2) was computed as: {[(Number of partial seizures per week at Baseline) minus (Number of partial seizures per week at Study Visit 4)] divided by (Number of partial seizures per week at Baseline)} multiplied by 100. A positive value in percent difference from Baseline indicates a reduction in partial seizure frequency from Baseline. Data of this outcome measure was analyzed and reported for participants on adjunctive therapy.
Time Frame: From Baseline (Week 0) to Visit 4 (up to Week 2)
Population: The FAS_A consisted of all participants in the SS_A who had at least 1 post-Baseline efficacy assessment.
Measure: Median (Full Range); unit: percent change
Arm/Group | Levetiracetam: Adjunctive Therapy
Number analyzed (Participants) | 32
percent change | 8.62 [-343.1 to 100.0]

3. Secondary Outcome: Percent Change in Partial Seizure Frequency Per Week From Baseline to Visit 5
Description: The percent difference in partial seizure frequency per week at Baseline and Study Visit 5 (Week 4) was computed as: {[(Number of partial seizures per week at Baseline) minus (Number of partial seizures per week at Study Visit 5)] divided by (Number of partial seizures per week at Baseline)} multiplied by 100. A positive value in percent difference from Baseline indicates a reduction in partial seizure frequency from Baseline. Data of this outcome measure was analyzed and reported for participants on adjunctive therapy.
Time Frame: From Baseline (Week 0) to Visit 5 (up to Week 4)
Population: The FAS_A consisted of all participants in the SS_A who had at least 1 post-Baseline efficacy assessment.
Measure: Median (Full Range); unit: percent change
Arm/Group | Levetiracetam: Adjunctive Therapy
Number analyzed (Participants) | 32
percent change | 16.79 [-414.3 to 100.0]

4. Secondary Outcome: Percent Change From Baseline for Each Analysis Visit in Partial Seizure Frequency Per Week on Adjunctive Therapy
Description: Percent difference in partial seizure frequency (PSF) per week at each Analysis Visit: {[(Number of partial seizures per week at Baseline [BL]) - (Number of partial seizures per week at analysis visit X)]/(Number of partial seizures per week at BL)}*100. Positive value indicates reduction in PSF from BL. End of study (EOS)/early discontinuation visit (EDV) was based on last EDV and calculation of number of partial seizure per week were based on the period from the previous EDV visit. The mapping of seizure data to Analysis Visits was based on target dates of the visits. A seizure date after that of target date of an Analysis Visit n and up to that of target date of next Analysis Visit n+1 was mapped to the next Analysis Visit (n+1). Data for one participant assessed within study duration was mapped to Analysis Visit 35/Week 300 based on statistical plan.
Time Frame: From Baseline (Week 0), Week 8, 10, 12, 15, 18, 21, 24, 27, 30, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, 192, 204, 216, 228, 240, 252, 264, 276, 288, 300, EOS/EDV (up to Week 295), and Safety follow-up (up to Week 295)
Population: The FAS_A consisted of all participants in the SS_A who had at least 1 post-Baseline efficacy assessment. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure. Here, number analyzed signifies participants who were evaluable at specified time points.
Measure: Median (Full Range); unit: percent change
Arm/Group | Levetiracetam: Adjunctive Therapy
Number analyzed (Participants) | 25
percent change
  Week 8 | 35.53 [-137.9 to 100.0]
  Week 10: number analyzed (Participants) | 24
  Week 10 | 59.39 [-138.2 to 100.0]
  Week 12: number analyzed (Participants) | 22
  Week 12 | 50.90 [-167.8 to 100.0]
  Week 15: number analyzed (Participants) | 22
  Week 15 | 60.29 [-129.4 to 100.0]
  Week 18: number analyzed (Participants) | 20
  Week 18 | 82.74 [-22.3 to 100.0]
  Week 21: number analyzed (Participants) | 20
  Week 21 | 80.33 [-44.1 to 100.0]
  Week 24: number analyzed (Participants) | 19
  Week 24 | 88.44 [-97.8 to 100.0]
  Week 27: number analyzed (Participants) | 18
  Week 27 | 93.84 [-4.8 to 100.0]
  Week 30: number analyzed (Participants) | 17
  Week 30 | 98.05 [-4.8 to 100.0]
  Week 36: number analyzed (Participants) | 16
  Week 36 | 100.00 [-94.5 to 100.0]
  Week 48: number analyzed (Participants) | 16
  Week 48 | 98.70 [-28.4 to 100.0]
  Week 60: number analyzed (Participants) | 13
  Week 60 | 100.00 [44.7 to 100.0]
  Week 72: number analyzed (Participants) | 13
  Week 72 | 100.00 [32.0 to 100.0]
  Week 84: number analyzed (Participants) | 13
  Week 84 | 100.00 [62.9 to 100.0]
  Week 96: number analyzed (Participants) | 12
  Week 96 | 99.57 [78.2 to 100.0]
  Week 108: number analyzed (Participants) | 11
  Week 108 | 100.00 [-48.0 to 100.0]
  Week 120: number analyzed (Participants) | 10
  Week 120 | 100.00 [80.4 to 100.0]
  Week 132: number analyzed (Participants) | 8
  Week 132 | 100.00 [50.7 to 100.0]
  Week 144: number analyzed (Participants) | 7
  Week 144 | 100.00 [93.4 to 100.0]
  Week 156: number analyzed (Participants) | 6
  Week 156 | 99.76 [93.5 to 100.0]
  Week 168: number analyzed (Participants) | 6
  Week 168 | 99.74 [90.7 to 100.0]
  Week 180: number analyzed (Participants) | 6
  Week 180 | 99.02 [86.1 to 100.0]
  Week 192: number analyzed (Participants) | 6
  Week 192 | 99.76 [85.5 to 100.0]
  Week 204: number analyzed (Participants) | 5
  Week 204 | 97.94 [78.3 to 100.0]
  Week 216: number analyzed (Participants) | 5
  Week 216 | 96.58 [81.4 to 100.0]
  Week 228: number analyzed (Participants) | 3
  Week 228 | 97.12 [96.6 to 100.0]
  Week 240: number analyzed (Participants) | 3
  Week 240 | 96.36 [86.8 to 100.0]
  Week 252: number analyzed (Participants) | 2
  Week 252 | 91.12 [85.3 to 96.9]
  Week 264: number analyzed (Participants) | 2
  Week 264 | 96.91 [95.8 to 98.0]
  Week 276: number analyzed (Participants) | 2
  Week 276 | 96.40 [95.2 to 97.6]
  Week 288: number analyzed (Participants) | 2
  Week 288 | 96.14 [94.2 to 98.0]
  Week 300: number analyzed (Participants) | 1
  Week 300 | 89.7 [89.7 to 89.7]
  EOS/EDV: number analyzed (Participants) | 10
  EOS/EDV | 21.86 [-120.1 to 100.0]
  Safety Follow Up: number analyzed (Participants) | 24
  Safety Follow Up | 39.82 [-267.8 to 100.0]

5. Secondary Outcome: Percentage of Participants With a Percent Change in Partial Seizure Frequency Per Week of <0%, 0% to <25%, 25% to <50%, ≥50%, ≥75%, or 100% on Adjunctive Therapy
Description: Percent difference in PSF per week on adjunctive therapy at BL and each analysis visit: {[(Number of partial seizures per week at BL) - (Number of partial seizures per week at analysis visit X)]/(Number of partial seizures per week at BL)}*100. Percent difference in PSF per week from Baseline for each participant and analysis visit were mapped into 6 categories: <0%, 0% to <25%, 25% to <50%, ≥50%, ≥75%, and 100%, then percentages of participants in these categories were derived using the number of participants at risk at each previous analysis visit as denominator. Positive value in percent difference from Baseline indicates reduction in PSF from Baseline. The mapping of seizure data to Analysis Visits was based on target dates of visits. A seizure date after that of target date of an Analysis Visit n and up to that of target date of next Analysis Visit n+1 was mapped to next Analysis Visit (n+1).
Time Frame: From Baseline (Week 0), Week 2, 4, 6, 8, 10, 12, 15, 18, 21, 24, 27, 30, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, 192, 204, 216, 228, 240, 252, 264, 276, 288, 300, EOS/EDV Week 2, EOS/EDV Week 4, and Safety follow-up (up to Week 295)
Population: FAS_A consisted of all participants in SS_A who had at least 1 post-Baseline efficacy assessment. Here, number analyzed signifies participants who were at risk at each previous analysis visit (X-1). As per planned analysis, outcome categories "≥50%", "≥75%" and "100%" are overlapping, so that percentages of categories of this outcome measure can add up to more than 100%. Data for one participant assessed within study duration was mapped to Analysis Visit 35/Week 300 based on statistical plan.
Measure: Number; unit: percentage of participants
Arm/Group | Levetiracetam: Adjunctive Therapy
Number analyzed (Participants) | 32
percentage of participants
  Week 2: <0% | 43.8
  Week 2: 0% - <25% | 18.8
  Week 2: 25% - <50% | 9.4
  Week 2: ≥ 50% | 28.1
  Week 2: ≥ 75% | 12.5
  Week 2: 100% | 9.4
  Week 4: <0% | 37.5
  Week 4: 0% - <25% | 18.8
  Week 4: 25% - <50% | 15.6
  Week 4: ≥ 50% | 28.1
  Week 4: ≥ 75% | 18.8
  Week 4: 100% | 9.4
  Week 6: <0% | 31.3
  Week 6: 0% - <25% | 15.6
  Week 6: 25% - <50% | 12.5
  Week 6: ≥ 50% | 28.1
  Week 6: ≥ 75% | 18.8
  Week 6: 100% | 15.6
  Week 8: <0%: number analyzed (Participants) | 28
  Week 8: <0% | 21.4
  Week 8: 0% - <25%: number analyzed (Participants) | 28
  Week 8: 0% - <25% | 14.3
  Week 8: 25% - <50%: number analyzed (Participants) | 28
  Week 8: 25% - <50% | 17.9
  Week 8: ≥ 50%: number analyzed (Participants) | 28
  Week 8: ≥ 50% | 35.7
  Week 8: ≥ 75%: number analyzed (Participants) | 28
  Week 8: ≥ 75% | 25.0
  Week 8: 100%: number analyzed (Participants) | 28
  Week 8: 100% | 17.9
  Week 10: <0%: number analyzed (Participants) | 25
  Week 10: <0% | 24.0
  Week 10: 0% - <25%: number analyzed (Participants) | 25
  Week 10: 0% - <25% | 12.0
  Week 10: 25% - <50%: number analyzed (Participants) | 25
  Week 10: 25% - <50% | 8.0
  Week 10: ≥ 50%: number analyzed (Participants) | 25
  Week 10: ≥ 50% | 52.0
  Week 10: ≥ 75%: number analyzed (Participants) | 25
  Week 10: ≥ 75% | 28.0
  Week 10: 100%: number analyzed (Participants) | 25
  Week 10: 100% | 20.0
  Week 12: <0%: number analyzed (Participants) | 24
  Week 12: <0% | 20.8
  Week 12: 0% - <25%: number analyzed (Participants) | 24
  Week 12: 0% - <25% | 4.2
  Week 12: 25% - <50%: number analyzed (Participants) | 24
  Week 12: 25% - <50% | 20.8
  Week 12: ≥ 50%: number analyzed (Participants) | 24
  Week 12: ≥ 50% | 45.8
  Week 12: ≥ 75%: number analyzed (Participants) | 24
  Week 12: ≥ 75% | 37.5
  Week 12: 100%: number analyzed (Participants) | 24
  Week 12: 100% | 25.0
  Week 15: <0%: number analyzed (Participants) | 22
  Week 15: <0% | 13.6
  Week 15: 0% - <25%: number analyzed (Participants) | 22
  Week 15: 0% - <25% | 9.1
  Week 15: 25% - <50%: number analyzed (Participants) | 22
  Week 15: 25% - <50% | 13.6
  Week 15: ≥ 50%: number analyzed (Participants) | 22
  Week 15: ≥ 50% | 63.6
  Week 15: ≥ 75%: number analyzed (Participants) | 22
  Week 15: ≥ 75% | 36.4
  Week 15: 100%: number analyzed (Participants) | 22
  Week 15: 100% | 27.3
  Week 18: <0%: number analyzed (Participants) | 22
  Week 18: <0% | 9.1
  Week 18: 0% - <25%: number analyzed (Participants) | 22
  Week 18: 0% - <25% | 4.5
  Week 18: 25% - <50%: number analyzed (Participants) | 22
  Week 18: 25% - <50% | 9.1
  Week 18: ≥ 50%: number analyzed (Participants) | 22
  Week 18: ≥ 50% | 68.2
  Week 18: ≥ 75%: number analyzed (Participants) | 22
  Week 18: ≥ 75% | 54.5
  Week 18: 100%: number analyzed (Participants) | 22
  Week 18: 100% | 31.8
  Week 21: <0%: number analyzed (Participants) | 20
  Week 21: <0% | 10.0
  Week 21: 0% - <25%: number analyzed (Participants) | 20
  Week 21: 0% - <25% | 5.0
  Week 21: 25% - <50%: number analyzed (Participants) | 20
  Week 21: 25% - <50% | 5.0
  Week 21: ≥ 50%: number analyzed (Participants) | 20
  Week 21: ≥ 50% | 80.0
  Week 21: ≥ 75%: number analyzed (Participants) | 20
  Week 21: ≥ 75% | 55.0
  Week 21: 100%: number analyzed (Participants) | 20
  Week 21: 100% | 30.0
  Week 24: <0%: number analyzed (Participants) | 20
  Week 24: <0% | 10.0
  Week 24: 0% - <25%: number analyzed (Participants) | 20
  Week 24: 0% - <25% | 10.0
  Week 24: 25% - <50%: number analyzed (Participants) | 20
  Week 24: 25% - <50% | 5.0
  Week 24: ≥ 50%: number analyzed (Participants) | 20
  Week 24: ≥ 50% | 70.0
  Week 24: ≥ 75%: number analyzed (Participants) | 20
  Week 24: ≥ 75% | 55.0
  Week 24: 100%: number analyzed (Participants) | 20
  Week 24: 100% | 40.0
  Week 27: <0%: number analyzed (Participants) | 19
  Week 27: <0% | 5.3
  Week 27: 0% - <25%: number analyzed (Participants) | 19
  Week 27: 0% - <25% | 5.3
  Week 27: 25% - <50%: number analyzed (Participants) | 19
  Week 27: 25% - <50% | 10.5
  Week 27: ≥ 50%: number analyzed (Participants) | 19
  Week 27: ≥ 50% | 73.7
  Week 27: ≥ 75%: number analyzed (Participants) | 19
  Week 27: ≥ 75% | 52.6
  Week 27: 100%: number analyzed (Participants) | 19
  Week 27: 100% | 36.8
  Week 30: <0%: number analyzed (Participants) | 18
  Week 30: <0% | 5.6
  Week 30: 0% - <25%: number analyzed (Participants) | 18
  Week 30: 0% - <25% | 11.1
  Week 30: 25% - <50%: number analyzed (Participants) | 18
  Week 30: 25% - <50% | 5.6
  Week 30: ≥ 50%: number analyzed (Participants) | 18
  Week 30: ≥ 50% | 72.2
  Week 30: ≥ 75%: number analyzed (Participants) | 18
  Week 30: ≥ 75% | 55.6
  Week 30: 100%: number analyzed (Participants) | 18
  Week 30: 100% | 44.4
  Week 36: <0%: number analyzed (Participants) | 17
  Week 36: <0% | 11.8
  Week 36: 0% - <25%: number analyzed (Participants) | 17
  Week 36: 0% - <25% | 5.9
  Week 36: 25% - <50%: number analyzed (Participants) | 17
  Week 36: 25% - <50% | 0
  Week 36: ≥ 50%: number analyzed (Participants) | 17
  Week 36: ≥ 50% | 76.5
  Week 36: ≥ 75%: number analyzed (Participants) | 17
  Week 36: ≥ 75% | 70.6
  Week 36: 100%: number analyzed (Participants) | 17
  Week 36: 100% | 52.9
  Week 48: <0%: number analyzed (Participants) | 16
  Week 48: <0% | 6.3
  Week 48: 0% - <25%: number analyzed (Participants) | 16
  Week 48: 0% - <25% | 12.5
  Week 48: 25% - <50%: number analyzed (Participants) | 16
  Week 48: 25% - <50% | 6.3
  Week 48: ≥ 50%: number analyzed (Participants) | 16
  Week 48: ≥ 50% | 75.0
  Week 48: ≥ 75%: number analyzed (Participants) | 16
  Week 48: ≥ 75% | 75.0
  Week 48:100%: number analyzed (Participants) | 16
  Week 48:100% | 43.8
  Week 60: <0%: number analyzed (Participants) | 16
  Week 60: <0% | 0
  Week 60: 0% - <25%: number analyzed (Participants) | 16
  Week 60: 0% - <25% | 0
  Week 60: 25% - <50%: number analyzed (Participants) | 16
  Week 60: 25% - <50% | 6.3
  Week 60: ≥ 50%: number analyzed (Participants) | 16
  Week 60: ≥ 50% | 75.0
  Week 60: ≥ 75%: number analyzed (Participants) | 16
  Week 60: ≥ 75% | 68.8
  Week 60: 100%: number analyzed (Participants) | 16
  Week 60: 100% | 43.8
  Week 72: <0%: number analyzed (Participants) | 13
  Week 72: <0% | 0
  Week 72: 0% - <25%: number analyzed (Participants) | 13
  Week 72: 0% - <25% | 0
  Week 72: 25% - <50%: number analyzed (Participants) | 13
  Week 72: 25% - <50% | 7.7
  Week 72: ≥ 50%: number analyzed (Participants) | 13
  Week 72: ≥ 50% | 92.3
  Week 72: ≥ 75%: number analyzed (Participants) | 13
  Week 72: ≥ 75% | 76.9
  Week 72: 100%: number analyzed (Participants) | 13
  Week 72: 100% | 53.8
  Week 84: <0%: number analyzed (Participants) | 13
  Week 84: <0% | 0
  Week 84: 0% - <25%: number analyzed (Participants) | 13
  Week 84: 0% - <25% | 0
  Week 84: 25% - <50%: number analyzed (Participants) | 13
  Week 84: 25% - <50% | 0
  Week 84: ≥ 50%: number analyzed (Participants) | 13
  Week 84: ≥ 50% | 100
  Week 84: ≥ 75%: number analyzed (Participants) | 13
  Week 84: ≥ 75% | 84.6
  Week 84: 100%: number analyzed (Participants) | 13
  Week 84: 100% | 53.8
  Week 96: <0%: number analyzed (Participants) | 13
  Week 96: <0% | 0
  Week 96: 0% - <25%: number analyzed (Participants) | 13
  Week 96: 0% - <25% | 0
  Week 96: 25% - <50%: number analyzed (Participants) | 13
  Week 96: 25% - <50% | 0
  Week 96: ≥ 50%: number analyzed (Participants) | 13
  Week 96: ≥ 50% | 92.3
  Week 96: ≥ 75%: number analyzed (Participants) | 13
  Week 96: ≥ 75% | 92.3
  Week 96: 100%: number analyzed (Participants) | 13
  Week 96: 100% | 46.2
  Week 108: <0%: number analyzed (Participants) | 12
  Week 108: <0% | 8.3
  Week 108: 0% - <25%: number analyzed (Participants) | 12
  Week 108: 0% - <25% | 0
  Week 108: 25% - <50%: number analyzed (Participants) | 12
  Week 108: 25% - <50% | 0
  Week 108: ≥ 50%: number analyzed (Participants) | 12
  Week 108: ≥ 50% | 83.3
  Week 108: ≥ 75%: number analyzed (Participants) | 12
  Week 108: ≥ 75% | 75.0
  Week 108: 100%: number analyzed (Participants) | 12
  Week 108: 100% | 50.0
  Week 120: <0%: number analyzed (Participants) | 11
  Week 120: <0% | 0
  Week 120: 0% - <25%: number analyzed (Participants) | 11
  Week 120: 0% - <25% | 0
  Week 120: 25% - <50%: number analyzed (Participants) | 11
  Week 120: 25% - <50% | 0
  Week 120: ≥ 50%: number analyzed (Participants) | 11
  Week 120: ≥ 50% | 90.9
  Week 120: ≥ 75%: number analyzed (Participants) | 11
  Week 120: ≥ 75% | 90.9
  Week 120: 100%: number analyzed (Participants) | 11
  Week 120: 100% | 63.6
  Week 132: <0%: number analyzed (Participants) | 10
  Week 132: <0% | 0
  Week 132: 0% - <25%: number analyzed (Participants) | 10
  Week 132: 0% - <25% | 0
  Week 132: 25% - <50%: number analyzed (Participants) | 10
  Week 132: 25% - <50% | 0
  Week 132: ≥ 50%: number analyzed (Participants) | 10
  Week 132: ≥ 50% | 80.0
  Week 132: ≥ 75%: number analyzed (Participants) | 10
  Week 132: ≥ 75% | 70.0
  Week 132: 100%: number analyzed (Participants) | 10
  Week 132: 100% | 50.0
  Week 144: <0%: number analyzed (Participants) | 8
  Week 144: <0% | 0
  Week 144: 0% - <25%: number analyzed (Participants) | 8
  Week 144: 0% - <25% | 0
  Week 144: 25% - <50%: number analyzed (Participants) | 8
  Week 144: 25% - <50% | 0
  Week 144: ≥ 50%: number analyzed (Participants) | 8
  Week 144: ≥ 50% | 87.5
  Week 144: ≥ 75%: number analyzed (Participants) | 8
  Week 144: ≥ 75% | 87.5
  Week 144: 100%: number analyzed (Participants) | 8
  Week 144: 100% | 50.0
  Week 156: <0%: number analyzed (Participants) | 7
  Week 156: <0% | 0
  Week 156: 0% - <25%: number analyzed (Participants) | 7
  Week 156: 0% - <25% | 0
  Week 156: 25% - <50%: number analyzed (Participants) | 7
  Week 156: 25% - <50% | 0
  Week 156: ≥ 50%: number analyzed (Participants) | 7
  Week 156: ≥ 50% | 85.7
  Week 156: ≥ 75%: number analyzed (Participants) | 7
  Week 156: ≥ 75% | 85.7
  Week 156: 100%: number analyzed (Participants) | 7
  Week 156: 100% | 42.9
  Week 168: <0%: number analyzed (Participants) | 6
  Week 168: <0% | 0
  Week 168: 0% - <25%: number analyzed (Participants) | 6
  Week 168: 0% - <25% | 0
  Week 168: 25% - <50%: number analyzed (Participants) | 6
  Week 168: 25% - <50% | 0
  Week 168: ≥ 50%: number analyzed (Participants) | 6
  Week 168: ≥ 50% | 100
  Week 168: ≥ 75%: number analyzed (Participants) | 6
  Week 168: ≥ 75% | 100
  Week 168: 100%: number analyzed (Participants) | 6
  Week 168: 100% | 50.0
  Week 180: <0%: number analyzed (Participants) | 6
  Week 180: <0% | 0
  Week 180: 0% - <25%: number analyzed (Participants) | 6
  Week 180: 0% - <25% | 0
  Week 180: 25% - <50%: number analyzed (Participants) | 6
  Week 180: 25% - <50% | 0
  Week 180: ≥ 50%: number analyzed (Participants) | 6
  Week 180: ≥ 50% | 100
  Week 180: ≥ 75%: number analyzed (Participants) | 6
  Week 180: ≥ 75% | 100
  Week 180: 100%: number analyzed (Participants) | 6
  Week 180: 100% | 50.0
  Week 192: <0%: number analyzed (Participants) | 6
  Week 192: <0% | 0
  Week 192: 0% - <25%: number analyzed (Participants) | 6
  Week 192: 0% - <25% | 0
  Week 192: 25% - <50%: number analyzed (Participants) | 6
  Week 192: 25% - <50% | 0
  Week 192: ≥ 50%: number analyzed (Participants) | 6
  Week 192: ≥ 50% | 100
  Week 192: ≥ 75%: number analyzed (Participants) | 6
  Week 192: ≥ 75% | 100
  Week 192: 100%: number analyzed (Participants) | 6
  Week 192: 100% | 50.0
  Week 204: <0%: number analyzed (Participants) | 6
  Week 204: <0% | 0
  Week 204: 0% - <25%: number analyzed (Participants) | 6
  Week 204: 0% - <25% | 0
  Week 204: 25% - <50%: number analyzed (Participants) | 6
  Week 204: 25% - <50% | 0
  Week 204: ≥ 50%: number analyzed (Participants) | 6
  Week 204: ≥ 50% | 83.3
  Week 204: ≥ 75%: number analyzed (Participants) | 6
  Week 204: ≥ 75% | 83.3
  Week 204: 100%: number analyzed (Participants) | 6
  Week 204: 100% | 16.7
  Week 216: <0%: number analyzed (Participants) | 5
  Week 216: <0% | 0
  Week 216: 0% - <25%: number analyzed (Participants) | 5
  Week 216: 0% - <25% | 0
  Week 216: 25% - <50%: number analyzed (Participants) | 5
  Week 216: 25% - <50% | 0
  Week 216: ≥ 50%: number analyzed (Participants) | 5
  Week 216: ≥ 50% | 100
  Week 216: ≥ 75%: number analyzed (Participants) | 5
  Week 216: ≥ 75% | 100
  Week 216: 100%: number analyzed (Participants) | 5
  Week 216: 100% | 20.0
  Week 228: <0%: number analyzed (Participants) | 5
  Week 228: <0% | 0
  Week 228: 0% - <25%: number analyzed (Participants) | 5
  Week 228: 0% - <25% | 0
  Week 228: 25% - <50%: number analyzed (Participants) | 5
  Week 228: 25% - <50% | 0
  Week 228: ≥ 50%: number analyzed (Participants) | 5
  Week 228: ≥ 50% | 60.0
  Week 228: ≥ 75%: number analyzed (Participants) | 5
  Week 228: ≥ 75% | 60.0
  Week 228: 100%: number analyzed (Participants) | 5
  Week 228: 100% | 20.0
  Week 240: <0%: number analyzed (Participants) | 3
  Week 240: <0% | 0
  Week 240: 0% - <25%: number analyzed (Participants) | 3
  Week 240: 0% - <25% | 0
  Week 240: 25% - <50%: number analyzed (Participants) | 3
  Week 240: 25% - <50% | 0
  Week 240: ≥ 50%: number analyzed (Participants) | 3
  Week 240: ≥ 50% | 100
  Week 240: ≥ 75%: number analyzed (Participants) | 3
  Week 240: ≥ 75% | 100
  Week 240: 100%: number analyzed (Participants) | 3
  Week 240: 100% | 33.3
  Week 252: <0%: number analyzed (Participants) | 3
  Week 252: <0% | 0
  Week 252: 0% - <25%: number analyzed (Participants) | 3
  Week 252: 0% - <25% | 0
  Week 252: 25% - <50%: number analyzed (Participants) | 3
  Week 252: 25% - <50% | 0
  Week 252: ≥ 50%: number analyzed (Participants) | 3
  Week 252: ≥ 50% | 66.7
  Week 252: ≥ 75%: number analyzed (Participants) | 3
  Week 252: ≥ 75% | 66.7
  Week 252: 100%: number analyzed (Participants) | 3
  Week 252: 100% | 0
  Week 264: <0%: number analyzed (Participants) | 2
  Week 264: <0% | 0
  Week 264: 0% - <25%: number analyzed (Participants) | 2
  Week 264: 0% - <25% | 0
  Week 264: 25% - <50%: number analyzed (Participants) | 2
  Week 264: 25% - <50% | 0
  Week 264: ≥ 50%: number analyzed (Participants) | 2
  Week 264: ≥ 50% | 100
  Week 264: ≥ 75%: number analyzed (Participants) | 2
  Week 264: ≥ 75% | 100
  Week 264: 100%: number analyzed (Participants) | 2
  Week 264: 100% | 0
  Week 276: <0%: number analyzed (Participants) | 2
  Week 276: <0% | 0
  Week 276: 0% - <25%: number analyzed (Participants) | 2
  Week 276: 0% - <25% | 0
  Week 276: 25% - <50%: number analyzed (Participants) | 2
  Week 276: 25% - <50% | 0
  Week 276: ≥ 50%: number analyzed (Participants) | 2
  Week 276: ≥ 50% | 100
  Week 276: ≥ 75%: number analyzed (Participants) | 2
  Week 276: ≥ 75% | 100
  Week 276: 100%: number analyzed (Participants) | 2
  Week 276: 100% | 0
  Week 288: <0%: number analyzed (Participants) | 2
  Week 288: <0% | 0
  Week 288: 0% - <25%: number analyzed (Participants) | 2
  Week 288: 0% - <25% | 0
  Week 288: 25% - <50%: number analyzed (Participants) | 2
  Week 288: 25% - <50% | 0
  Week 288: ≥ 50%: number analyzed (Participants) | 2
  Week 288: ≥ 50% | 100
  Week 288: ≥ 75%: number analyzed (Participants) | 2
  Week 288: ≥ 75% | 100
  Week 288: 100%: number analyzed (Participants) | 2
  Week 288: 100% | 0
  Week 300: <0%: number analyzed (Participants) | 2
  Week 300: <0% | 0
  Week 300: 0% - <25%: number analyzed (Participants) | 2
  Week 300: 0% - <25% | 0
  Week 300: 25% - <50%: number analyzed (Participants) | 2
  Week 300: 25% - <50% | 0
  Week 300: ≥ 50%: number analyzed (Participants) | 2
  Week 300: ≥ 50% | 50.0
  Week 300: ≥ 75%: number analyzed (Participants) | 2
  Week 300: ≥ 75% | 50.0
  Week 300: 100%: number analyzed (Participants) | 2
  Week 300: 100% | 0
  EOS/EDV, Week 2: <0% | 3.1
  EOS/EDV, Week 2: 0% - <25% | 3.1
  EOS/EDV, Week 2: 25% - <50% | 0
  EOS/EDV, Week 2: ≥ 50% | 3.1
  EOS/EDV, Week 2: ≥ 75% | 3.1
  EOS/EDV, Week 2: 100% | 3.1
  EOS/EDV, Week 4: <0%: number analyzed (Participants) | 10
  EOS/EDV, Week 4: <0% | 20.0
  EOS/EDV, Week 4: 0% - <25%: number analyzed (Participants) | 10
  EOS/EDV, Week 4: 0% - <25% | 10.0
  EOS/EDV, Week 4: 25% - <50%: number analyzed (Participants) | 10
  EOS/EDV, Week 4: 25% - <50% | 20.0
  EOS/EDV, Week 4: ≥ 50%: number analyzed (Participants) | 10
  EOS/EDV, Week 4: ≥ 50% | 20.0
  EOS/EDV, Week 4: ≥ 75%: number analyzed (Participants) | 10
  EOS/EDV, Week 4: ≥ 75% | 10.0
  EOS/EDV, Week 4: 100%: number analyzed (Participants) | 10
  EOS/EDV, Week 4: 100% | 0
  Safety Follow Up: <0%: number analyzed (Participants) | 24
  Safety Follow Up: <0% | 37.5
  Safety Follow Up: 0% - <25%: number analyzed (Participants) | 24
  Safety Follow Up: 0% - <25% | 4.2
  Safety Follow Up: 25% - <50%: number analyzed (Participants) | 24
  Safety Follow Up: 25% - <50% | 12.5
  Safety Follow Up: ≥ 50%: number analyzed (Participants) | 24
  Safety Follow Up: ≥ 50% | 45.8
  Safety Follow Up: ≥ 75%: number analyzed (Participants) | 24
  Safety Follow Up: ≥ 75% | 29.2
  Safety Follow Up: 100%: number analyzed (Participants) | 24
  Safety Follow Up: 100% | 20.8

6. Secondary Outcome: Percent Change From Baseline for Each Analysis Visit in Partial Seizure Frequency Per Week on Monotherapy
Description: The percent difference in partial seizure frequency per week on monotherapy at Baseline and each analysis visit was computed as: {[(Number of partial seizures per week at Baseline) minus (Number of partial seizures per week at analysis visit X)] divided by (Number of partial seizures per week at Baseline)} multiplied by 100. A positive value in percent difference from Baseline indicates a reduction in partial seizure frequency from Baseline. Data of this outcome measure was analyzed and reported for participants on monotherapy. The maximum duration of study participation in monotherapy participants was shorter than in adjunctive therapy. Therefore, data at Week 288 and 300 is not reported for Monotherapy.
Time Frame: From Baseline (Week 0), Week 2, 4, 6, 8, 10, 12, 15, 18, 21, 24, 27, 30, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, 192, 204, 216, 228, 240, 252, 264, 276, and Safety follow-up (up to Week 295)
Population: The FAS_M consisted of all participants in the SS_M who had at least 1 post-Baseline efficacy assessment. Here, number analyzed signifies participants who were evaluable at specified time points.
Measure: Median (Full Range); unit: percent change
Arm/Group | Levetiracetam: Monotherapy
Number analyzed (Participants) | 6
percent change
  Week 2 | -51.87 [-731.6 to 100.0]
  Week 4 | 4.88 [-115.9 to 100.0]
  Week 6 | 51.10 [-325.0 to 100.0]
  Week 8: number analyzed (Participants) | 5
  Week 8 | 100.00 [-1.1 to 100.0]
  Week 10: number analyzed (Participants) | 5
  Week 10 | 100.00 [-277.1 to 100.0]
  Week 12: number analyzed (Participants) | 5
  Week 12 | 76.92 [-10.0 to 100.0]
  Week 15: number analyzed (Participants) | 5
  Week 15 | 100.00 [-78.1 to 100.0]
  Week 18: number analyzed (Participants) | 5
  Week 18 | 91.58 [58.1 to 100.0]
  Week 21: number analyzed (Participants) | 5
  Week 21 | 100.00 [76.9 to 100.0]
  Week 24: number analyzed (Participants) | 5
  Week 24 | 100.00 [92.3 to 100.0]
  Week 27: number analyzed (Participants) | 5
  Week 27 | 100.00 [26.7 to 100.0]
  Week 30: number analyzed (Participants) | 5
  Week 30 | 100.00 [37.1 to 100.0]
  Week 36: number analyzed (Participants) | 5
  Week 36 | 100.00 [16.2 to 100.0]
  Week 48: number analyzed (Participants) | 5
  Week 48 | 98.08 [-138.3 to 100.0]
  Week 60: number analyzed (Participants) | 5
  Week 60 | 94.23 [-41.4 to 100.0]
  Week 72: number analyzed (Participants) | 5
  Week 72 | 92.31 [-36.2 to 100.0]
  Week 84: number analyzed (Participants) | 5
  Week 84 | 95.79 [-86.0 to 100.0]
  Week 96: number analyzed (Participants) | 5
  Week 96 | 98.08 [-65.0 to 100.0]
  Week 108: number analyzed (Participants) | 5
  Week 108 | 96.15 [-44.0 to 100.0]
  Week 120: number analyzed (Participants) | 5
  Week 120 | 93.68 [-46.7 to 100.0]
  Week 132: number analyzed (Participants) | 4
  Week 132 | 92.63 [-138.3 to 100.0]
  Week 144: number analyzed (Participants) | 4
  Week 144 | 92.63 [-106.9 to 100.0]
  Week 156: number analyzed (Participants) | 4
  Week 156 | 94.73 [8.3 to 100.0]
  Week 168: number analyzed (Participants) | 4
  Week 168 | 100.00 [-70.2 to 100.0]
  Week 180: number analyzed (Participants) | 3
  Week 180 | 100.00 [-274.5 to 100.0]
  Week 192: number analyzed (Participants) | 3
  Week 192 | 100.00 [-223.0 to 100.0]
  Week 204: number analyzed (Participants) | 2
  Week 204 | 100.00 [100.0 to 100.0]
  Week 216: number analyzed (Participants) | 2
  Week 216 | 100.00 [100.0 to 100.0]
  Week 228: number analyzed (Participants) | 1
  Week 228 | 100.00 [100.0 to 100.0]
  Week 240: number analyzed (Participants) | 1
  Week 240 | 100.00 [100.00 to 100.00]
  Week 252: number analyzed (Participants) | 1
  Week 252 | 100.00 [100.00 to 100.00]
  Week 264: number analyzed (Participants) | 1
  Week 264 | 100.00 [100.00 to 100.00]
  Week 276: number analyzed (Participants) | 1
  Week 276 | 100.00 [100.00 to 100.00]
  Safety Follow Up: number analyzed (Participants) | 2
  Safety Follow Up | 100.0 [100.0 to 100.0]

7. Secondary Outcome: Percentage of Participants With a Percent Change in Partial Seizure Frequency Per Week of <0%, 0% to <25%, 25% to <50%, ≥50%, ≥75%, or 100% on Monotherapy
Description: Percent difference in PSF per week on monotherapy at BL and each analysis visit: {[(Number of partial seizures per week at BL) - (Number of partial seizures per week at analysis visit X)]/(Number of partial seizures per week at BL)}*100. Percent difference in PFS per week from Baseline for each participant and analysis visit were mapped into 6 categories: <0%, 0% to <25%, 25% to <50%, ≥50%, ≥75%, and 100%, then percentages of participants in these categories were derived using the number of participants at risk at each previous analysis visit as denominator. A positive value in percent difference from Baseline indicates a reduction in partial seizure frequency from Baseline. Data of this outcome measure was analyzed and reported for participants on monotherapy. Maximum duration of study participation in monotherapy participants was shorter than adjunctive therapy. Therefore, data at Week 288 and 300 is not reported for Monotherapy.
Time Frame: as for outcome 6
Population: The FAS_M consisted of all participants in the SS_M who had at least 1 post-Baseline efficacy assessment. Here, number analyzed signifies participants who were at risk at each previous analysis visit (X-1). As per planned analysis, outcome categories "≥50%", "≥75%" and "100%" are overlapping, so that percentages of categories of this outcome measure can add up to more than 100%.
Measure: Number; unit: percentage of participants
Arm/Group | Levetiracetam: Monotherapy
Number analyzed (Participants) | 6
percentage of participants
  Week 2: <0%: number analyzed (Participants) | 5
  Week 2: <0% | 60.0
  Week 2: 0% - <25%: number analyzed (Participants) | 5
  Week 2: 0% - <25% | 0
  Week 2: 25% - <50%: number analyzed (Participants) | 5
  Week 2: 25% - <50% | 20.0
  Week 2: ≥ 50%: number analyzed (Participants) | 5
  Week 2: ≥ 50% | 40.0
  Week 2: ≥ 75%: number analyzed (Participants) | 5
  Week 2: ≥ 75% | 20.0
  Week 2: 100%: number analyzed (Participants) | 5
  Week 2: 100% | 20.0
  Week 4: <0% | 50.0
  Week 4: 0% - <25% | 0
  Week 4: 25% - <50% | 16.7
  Week 4: ≥ 50% | 33.3
  Week 4: ≥ 75% | 33.3
  Week 4: 100% | 33.3
  Week 6: <0% | 33.3
  Week 6: 0% - <25% | 0
  Week 6: 25% - <50% | 16.7
  Week 6: ≥ 50% | 50.0
  Week 6: ≥ 75% | 33.3
  Week 6: 100% | 16.7
  Week 8: <0% | 16.7
  Week 8: 0% - <25% | 16.7
  Week 8: 25% - <50% | 0
  Week 8: ≥ 50% | 50.0
  Week 8: ≥ 75% | 50.0
  Week 8: 100% | 50.0
  Week 10: <0%: number analyzed (Participants) | 5
  Week 10: <0% | 20.0
  Week 10: 0% - <25%: number analyzed (Participants) | 5
  Week 10: 0% - <25% | 0
  Week 10: 25% - <50%: number analyzed (Participants) | 5
  Week 10: 25% - <50% | 0
  Week 10: ≥ 50%: number analyzed (Participants) | 5
  Week 10: ≥ 50% | 80.0
  Week 10: ≥ 75%: number analyzed (Participants) | 5
  Week 10: ≥ 75% | 80.0
  Week 10: 100%: number analyzed (Participants) | 5
  Week 10: 100% | 60.0
  Week 12: <0%: number analyzed (Participants) | 5
  Week 12: <0% | 20.0
  Week 12: 0% - <25%: number analyzed (Participants) | 5
  Week 12: 0% - <25% | 0
  Week 12: 25% - <50%: number analyzed (Participants) | 5
  Week 12: 25% - <50% | 20.0
  Week 12: ≥ 50%: number analyzed (Participants) | 5
  Week 12: ≥ 50% | 60.0
  Week 12: ≥ 75%: number analyzed (Participants) | 5
  Week 12: ≥ 75% | 60.0
  Week 12: 100%: number analyzed (Participants) | 5
  Week 12: 100% | 40.0
  Week 15: <0%: number analyzed (Participants) | 5
  Week 15: <0% | 20.0
  Week 15: 0% - <25%: number analyzed (Participants) | 5
  Week 15: 0% - <25% | 0
  Week 15: 25% - <50%: number analyzed (Participants) | 5
  Week 15: 25% - <50% | 20.0
  Week 15: ≥ 50%: number analyzed (Participants) | 5
  Week 15: ≥ 50% | 60.0
  Week 15: ≥ 75%: number analyzed (Participants) | 5
  Week 15: ≥ 75% | 60.0
  Week 15: 100%: number analyzed (Participants) | 5
  Week 15: 100% | 60.0
  Week 18: <0%: number analyzed (Participants) | 5
  Week 18: <0% | 0
  Week 18: 0% - <25%: number analyzed (Participants) | 5
  Week 18: 0% - <25% | 0
  Week 18: 25% - <50%: number analyzed (Participants) | 5
  Week 18: 25% - <50% | 0
  Week 18: ≥ 50%: number analyzed (Participants) | 5
  Week 18: ≥ 50% | 100
  Week 18: ≥ 75%: number analyzed (Participants) | 5
  Week 18: ≥ 75% | 80.0
  Week 18: 100%: number analyzed (Participants) | 5
  Week 18: 100% | 40.0
  Week 21: <0%: number analyzed (Participants) | 5
  Week 21: <0% | 0
  Week 21: 0% - <25%: number analyzed (Participants) | 5
  Week 21: 0% - <25% | 0
  Week 21: 25% - <50%: number analyzed (Participants) | 5
  Week 21: 25% - <50% | 0
  Week 21: ≥ 50%: number analyzed (Participants) | 5
  Week 21: ≥ 50% | 100
  Week 21: ≥ 75%: number analyzed (Participants) | 5
  Week 21: ≥ 75% | 100
  Week 21: 100%: number analyzed (Participants) | 5
  Week 21: 100% | 60.0
  Week 24: <0%: number analyzed (Participants) | 5
  Week 24: <0% | 0
  Week 24: 0% - <25%: number analyzed (Participants) | 5
  Week 24: 0% - <25% | 0
  Week 24: 25% - <50%: number analyzed (Participants) | 5
  Week 24: 25% - <50% | 0
  Week 24: ≥ 50%: number analyzed (Participants) | 5
  Week 24: ≥ 50% | 100
  Week 24: ≥ 75%: number analyzed (Participants) | 5
  Week 24: ≥ 75% | 100
  Week 24: 100%: number analyzed (Participants) | 5
  Week 24: 100% | 80.0
  Week 27: <0%: number analyzed (Participants) | 5
  Week 27: <0% | 0
  Week 27: 0% - <25%: number analyzed (Participants) | 5
  Week 27: 0% - <25% | 0
  Week 27: 25% - <50%: number analyzed (Participants) | 5
  Week 27: 25% - <50% | 20.0
  Week 27: ≥ 50%: number analyzed (Participants) | 5
  Week 27: ≥ 50% | 80.0
  Week 27: ≥ 75%: number analyzed (Participants) | 5
  Week 27: ≥ 75% | 80.0
  Week 27: 100%: number analyzed (Participants) | 5
  Week 27: 100% | 80.0
  Week 30: <0%: number analyzed (Participants) | 5
  Week 30: <0% | 0
  Week 30: 0% - <25%: number analyzed (Participants) | 5
  Week 30: 0% - <25% | 0
  Week 30: 25% - <50%: number analyzed (Participants) | 5
  Week 30: 25% - <50% | 20.0
  Week 30: ≥ 50%: number analyzed (Participants) | 5
  Week 30: ≥ 50% | 80.0
  Week 30: ≥ 75%: number analyzed (Participants) | 5
  Week 30: ≥ 75% | 60.0
  Week 30: 100%: number analyzed (Participants) | 5
  Week 30: 100% | 60.0
  Week 36: <0%: number analyzed (Participants) | 5
  Week 36: <0% | 0
  Week 36: 0% - <25%: number analyzed (Participants) | 5
  Week 36: 0% - <25% | 20.0
  Week 36: 25% - <50%: number analyzed (Participants) | 5
  Week 36: 25% - <50% | 0
  Week 36: ≥ 50%: number analyzed (Participants) | 5
  Week 36: ≥ 50% | 80.0
  Week 36: ≥ 75%: number analyzed (Participants) | 5
  Week 36: ≥ 75% | 80.0
  Week 36: 100%: number analyzed (Participants) | 5
  Week 36: 100% | 60.0
  Week 48: <0%: number analyzed (Participants) | 5
  Week 48: <0% | 20.0
  Week 48: 0% - <25%: number analyzed (Participants) | 5
  Week 48: 0% - <25% | 0
  Week 48: 25% - <50%: number analyzed (Participants) | 5
  Week 48: 25% - <50% | 0
  Week 48: ≥ 50%: number analyzed (Participants) | 5
  Week 48: ≥ 50% | 80.0
  Week 48: ≥ 75%: number analyzed (Participants) | 5
  Week 48: ≥ 75% | 80.0
  Week 48:100%: number analyzed (Participants) | 5
  Week 48:100% | 40.0
  Week 60: <0%: number analyzed (Participants) | 5
  Week 60: <0% | 20.0
  Week 60: 0% - <25%: number analyzed (Participants) | 5
  Week 60: 0% - <25% | 0
  Week 60: 25% - <50%: number analyzed (Participants) | 5
  Week 60: 25% - <50% | 0
  Week 60: ≥ 50%: number analyzed (Participants) | 5
  Week 60: ≥ 50% | 80.0
  Week 60: ≥ 75%: number analyzed (Participants) | 5
  Week 60: ≥ 75% | 80.0
  Week 60: 100%: number analyzed (Participants) | 5
  Week 60: 100% | 40.0
  Week 72: <0%: number analyzed (Participants) | 5
  Week 72: <0% | 20.0
  Week 72: 0% - <25%: number analyzed (Participants) | 5
  Week 72: 0% - <25% | 0
  Week 72: 25% - <50%: number analyzed (Participants) | 5
  Week 72: 25% - <50% | 0
  Week 72: ≥ 50%: number analyzed (Participants) | 5
  Week 72: ≥ 50% | 80.0
  Week 72: ≥ 75%: number analyzed (Participants) | 5
  Week 72: ≥ 75% | 80.0
  Week 72: 100%: number analyzed (Participants) | 5
  Week 72: 100% | 40.0
  Week 84: <0%: number analyzed (Participants) | 5
  Week 84: <0% | 20.0
  Week 84: 0% - <25%: number analyzed (Participants) | 5
  Week 84: 0% - <25% | 0
  Week 84: 25% - <50%: number analyzed (Participants) | 5
  Week 84: 25% - <50% | 0
  Week 84: ≥ 50%: number analyzed (Participants) | 5
  Week 84: ≥ 50% | 80.0
  Week 84: ≥ 75%: number analyzed (Participants) | 5
  Week 84: ≥ 75% | 80.0
  Week 84: 100%: number analyzed (Participants) | 5
  Week 84: 100% | 40.0
  Week 96: <0%: number analyzed (Participants) | 5
  Week 96: <0% | 20.0
  Week 96: 0% - <25%: number analyzed (Participants) | 5
  Week 96: 0% - <25% | 0
  Week 96: 25% - <50%: number analyzed (Participants) | 5
  Week 96: 25% - <50% | 0
  Week 96: ≥ 50%: number analyzed (Participants) | 5
  Week 96: ≥ 50% | 80.0
  Week 96: ≥ 75%: number analyzed (Participants) | 5
  Week 96: ≥ 75% | 80.0
  Week 96: 100%: number analyzed (Participants) | 5
  Week 96: 100% | 40.0
  Week 108: <0%: number analyzed (Participants) | 5
  Week 108: <0% | 20.0
  Week 108: 0% - <25%: number analyzed (Participants) | 5
  Week 108: 0% - <25% | 0
  Week 108: 25% - <50%: number analyzed (Participants) | 5
  Week 108: 25% - <50% | 0
  Week 108: ≥ 50%: number analyzed (Participants) | 5
  Week 108: ≥ 50% | 80.0
  Week 108: ≥ 75%: number analyzed (Participants) | 5
  Week 108: ≥ 75% | 80.0
  Week 108: 100%: number analyzed (Participants) | 5
  Week 108: 100% | 40.0
  Week 120: <0%: number analyzed (Participants) | 5
  Week 120: <0% | 20.0
  Week 120: 0% - <25%: number analyzed (Participants) | 5
  Week 120: 0% - <25% | 0
  Week 120: 25% - <50%: number analyzed (Participants) | 5
  Week 120: 25% - <50% | 0
  Week 120: ≥ 50%: number analyzed (Participants) | 5
  Week 120: ≥ 50% | 80.0
  Week 120: ≥ 75%: number analyzed (Participants) | 5
  Week 120: ≥ 75% | 80.0
  Week 120: 100%: number analyzed (Participants) | 5
  Week 120: 100% | 40.0
  Week 132: <0%: number analyzed (Participants) | 5
  Week 132: <0% | 20.0
  Week 132: 0% - <25%: number analyzed (Participants) | 5
  Week 132: 0% - <25% | 0
  Week 132: 25% - <50%: number analyzed (Participants) | 5
  Week 132: 25% - <50% | 0
  Week 132: ≥ 50%: number analyzed (Participants) | 5
  Week 132: ≥ 50% | 60.0
  Week 132: ≥ 75%: number analyzed (Participants) | 5
  Week 132: ≥ 75% | 60.0
  Week 132: 100%: number analyzed (Participants) | 5
  Week 132: 100% | 40.0
  Week 144: <0%: number analyzed (Participants) | 4
  Week 144: <0% | 25.0
  Week 144: 0% - <25%: number analyzed (Participants) | 4
  Week 144: 0% - <25% | 0
  Week 144: 25% - <50%: number analyzed (Participants) | 4
  Week 144: 25% - <50% | 0
  Week 144: ≥ 50%: number analyzed (Participants) | 4
  Week 144: ≥ 50% | 75.0
  Week 144: ≥ 75%: number analyzed (Participants) | 4
  Week 144: ≥ 75% | 75.0
  Week 144: 100%: number analyzed (Participants) | 4
  Week 144: 100% | 50.0
  Week 156: <0%: number analyzed (Participants) | 4
  Week 156: <0% | 0
  Week 156: 0% - <25%: number analyzed (Participants) | 4
  Week 156: 0% - <25% | 25.0
  Week 156: 25% - <50%: number analyzed (Participants) | 4
  Week 156: 25% - <50% | 0
  Week 156: ≥ 50%: number analyzed (Participants) | 4
  Week 156: ≥ 50% | 75.0
  Week 156: ≥ 75%: number analyzed (Participants) | 4
  Week 156: ≥ 75% | 75.0
  Week 156: 100%: number analyzed (Participants) | 4
  Week 156: 100% | 50.0
  Week 168: <0%: number analyzed (Participants) | 4
  Week 168: <0% | 25.0
  Week 168: 0% - <25%: number analyzed (Participants) | 4
  Week 168: 0% - <25% | 0
  Week 168: 25% - <50%: number analyzed (Participants) | 4
  Week 168: 25% - <50% | 0
  Week 168: ≥ 50%: number analyzed (Participants) | 4
  Week 168: ≥ 50% | 75.0
  Week 168: ≥ 75%: number analyzed (Participants) | 4
  Week 168: ≥ 75% | 75.0
  Week 168: 100%: number analyzed (Participants) | 4
  Week 168: 100% | 75.0
  Week 180: <0%: number analyzed (Participants) | 4
  Week 180: <0% | 25.0
  Week 180: 0% - <25%: number analyzed (Participants) | 4
  Week 180: 0% - <25% | 0
  Week 180: 25% - <50%: number analyzed (Participants) | 4
  Week 180: 25% - <50% | 0
  Week 180: ≥ 50%: number analyzed (Participants) | 4
  Week 180: ≥ 50% | 50.0
  Week 180: ≥ 75%: number analyzed (Participants) | 4
  Week 180: ≥ 75% | 50.0
  Week 180: 100%: number analyzed (Participants) | 4
  Week 180: 100% | 50.0
  Week 192: <0%: number analyzed (Participants) | 3
  Week 192: <0% | 33.3
  Week 192: 0% - <25%: number analyzed (Participants) | 3
  Week 192: 0% - <25% | 0
  Week 192: 25% - <50%: number analyzed (Participants) | 3
  Week 192: 25% - <50% | 0
  Week 192: ≥ 50%: number analyzed (Participants) | 3
  Week 192: ≥ 50% | 66.7
  Week 192: ≥ 75%: number analyzed (Participants) | 3
  Week 192: ≥ 75% | 66.7
  Week 192: 100%: number analyzed (Participants) | 3
  Week 192: 100% | 66.7
  Week 204: <0%: number analyzed (Participants) | 3
  Week 204: <0% | 0
  Week 204: 0% - <25%: number analyzed (Participants) | 3
  Week 204: 0% - <25% | 0
  Week 204: 25% - <50%: number analyzed (Participants) | 3
  Week 204: 25% - <50% | 0
  Week 204: ≥ 50%: number analyzed (Participants) | 3
  Week 204: ≥ 50% | 66.7
  Week 204: ≥ 75%: number analyzed (Participants) | 3
  Week 204: ≥ 75% | 66.7
  Week 204: 100%: number analyzed (Participants) | 3
  Week 204: 100% | 66.7
  Week 216: <0%: number analyzed (Participants) | 2
  Week 216: <0% | 0
  Week 216: 0% - <25%: number analyzed (Participants) | 2
  Week 216: 0% - <25% | 0
  Week 216: 25% - <50%: number analyzed (Participants) | 2
  Week 216: 25% - <50% | 0
  Week 216: ≥ 50%: number analyzed (Participants) | 2
  Week 216: ≥ 50% | 100
  Week 216: ≥ 75%: number analyzed (Participants) | 2
  Week 216: ≥ 75% | 100
  Week 216: 100%: number analyzed (Participants) | 2
  Week 216: 100% | 100
  Week 228: <0%: number analyzed (Participants) | 2
  Week 228: <0% | 0
  Week 228: 0% - <25%: number analyzed (Participants) | 2
  Week 228: 0% - <25% | 0
  Week 228: 25% - <50%: number analyzed (Participants) | 2
  Week 228: 25% - <50% | 0
  Week 228: ≥ 50%: number analyzed (Participants) | 2
  Week 228: ≥ 50% | 50.0
  Week 228: ≥ 75%: number analyzed (Participants) | 2
  Week 228: ≥ 75% | 50.0
  Week 228: 100%: number analyzed (Participants) | 2
  Week 228: 100% | 50.0
  Week 240: <0%: number analyzed (Participants) | 1
  Week 240: <0% | 0
  Week 240: 0% - <25%: number analyzed (Participants) | 1
  Week 240: 0% - <25% | 0
  Week 240: 25% - <50%: number analyzed (Participants) | 1
  Week 240: 25% - <50% | 0
  Week 240: ≥ 50%: number analyzed (Participants) | 1
  Week 240: ≥ 50% | 100
  Week 240: ≥ 75%: number analyzed (Participants) | 1
  Week 240: ≥ 75% | 100
  Week 240: 100%: number analyzed (Participants) | 1
  Week 240: 100% | 100
  Week 252: <0%: number analyzed (Participants) | 1
  Week 252: <0% | 0
  Week 252: 0% - <25%: number analyzed (Participants) | 1
  Week 252: 0% - <25% | 0
  Week 252: 25% - <50%: number analyzed (Participants) | 1
  Week 252: 25% - <50% | 0
  Week 252: ≥ 50%: number analyzed (Participants) | 1
  Week 252: ≥ 50% | 100
  Week 252: ≥ 75%: number analyzed (Participants) | 1
  Week 252: ≥ 75% | 100
  Week 252: 100%: number analyzed (Participants) | 1
  Week 252: 100% | 100
  Week 264: <0%: number analyzed (Participants) | 1
  Week 264: <0% | 0
  Week 264: 0% - <25%: number analyzed (Participants) | 1
  Week 264: 0% - <25% | 0
  Week 264: 25% - <50%: number analyzed (Participants) | 1
  Week 264: 25% - <50% | 0
  Week 264: ≥ 50%: number analyzed (Participants) | 1
  Week 264: ≥ 50% | 100
  Week 264: ≥ 75%: number analyzed (Participants) | 1
  Week 264: ≥ 75% | 100
  Week 264: 100%: number analyzed (Participants) | 1
  Week 264: 100% | 100
  Week 276: <0%: number analyzed (Participants) | 1
  Week 276: <0% | 0
  Week 276: 0% - <25%: number analyzed (Participants) | 1
  Week 276: 0% - <25% | 0
  Week 276: 25% - <50%: number analyzed (Participants) | 1
  Week 276: 25% - <50% | 0
  Week 276: ≥ 50%: number analyzed (Participants) | 1
  Week 276: ≥ 50% | 100
  Week 276: ≥ 75%: number analyzed (Participants) | 1
  Week 276: ≥ 75% | 100
  Week 276: 100%: number analyzed (Participants) | 1
  Week 276: 100% | 100
  Safety Follow Up: <0%: number analyzed (Participants) | 2
  Safety Follow Up: <0% | 0
  Safety Follow Up: 0% - <25%: number analyzed (Participants) | 2
  Safety Follow Up: 0% - <25% | 0
  Safety Follow Up: 25% - <50%: number analyzed (Participants) | 2
  Safety Follow Up: 25% - <50% | 0
  Safety Follow Up: ≥ 50%: number analyzed (Participants) | 2
  Safety Follow Up: ≥ 50% | 100
  Safety Follow Up: ≥ 75%: number analyzed (Participants) | 2
  Safety Follow Up: ≥ 75% | 100
  Safety Follow Up: 100%: number analyzed (Participants) | 2
  Safety Follow Up: 100% | 100

8. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) During the First Period
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation Participant administered a pharmaceutical product that does not necessarily have a causal relationship treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. The treatment-emergent adverse events (TEAEs) were defined as those events that started on or after the date (and time) of first dose of study medication, or adverse events whose intensity worsened on or after the date (and time) of first dose of study medication.
Time Frame: From Baseline (Week 0) to Visit 6 (up to Week 6)
Population: The SS_A consisted of all enrolled participants on adjunctive therapy who received at least 1 dose of study medication in the evaluation period. The SS_M consisted of all enrolled participants on monotherapy who received at least 1 dose of study medication in the evaluation period.
Measure: Number; unit: percentage of participants
Arm/Group | Levetiracetam: Adjunctive Therapy | Levetiracetam: Monotherapy
Number analyzed (Participants) | 32 | 6
percentage of participants | 62.5 | 0

9. Secondary Outcome: Percentage of Participants With Treatment-emergent Serious Adverse Events (SAEs) During the First Period
Description: A serious adverse event (SAE) is defined as any untoward medical occurrence at any dose that must meet 1 or more of the following criteria: Death; Life-threatening; Significant or persistent disability/incapacity; Congenital anomaly/birth defect (including that occurring in a fetus); Important medical event that, based upon appropriate medical judgment, may jeopardize the patient or participant and may require medical or surgical intervention to prevent 1 of the other outcomes listed in the definition of serious; Initial inpatient hospitalization or prolongation of hospitalization. The TEAEs were defined as those events that started on or after the date (and time) of first dose of study medication, or adverse events whose intensity worsened on or after the date (and time) of first dose of study medication.
Time Frame: From Baseline (Week 0) to Visit 6 (up to Week 6)
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Levetiracetam: Adjunctive Therapy | Levetiracetam: Monotherapy
Number analyzed (Participants) | 32 | 6
percentage of participants | 9.4 | 0

10. Secondary Outcome: Percentage of Participants With TEAEs Leading to Discontinuation From Study Medication During the First Period
Description: An AE is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product that does not necessarily have a causal relationship treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. The TEAEs were defined as those events that started on or after the date (and time) of first dose of study medication, or adverse events whose intensity worsened on or after the date (and time) of first dose of study medication. TEAEs leading to discontinuation from study medication are reported.
Time Frame: From Baseline (Week 0) to Visit 6 (up to Week 6)
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Levetiracetam: Adjunctive Therapy | Levetiracetam: Monotherapy
Number analyzed (Participants) | 32 | 6
percentage of participants | 6.3 | 0

11. Secondary Outcome: Percentage of Participants With TEAEs During the Combined First and Second Period
Description: An AE is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product that does not necessarily have a causal relationship treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. The TEAEs were defined as those events that started on or after the date (and time) of first dose of study medication, or adverse events whose intensity worsened on or after the date (and time) of first dose of study medication.
Time Frame: From Baseline (Week 0) to the End of Safety Follow-up (up to Week 295)
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Levetiracetam: Adjunctive Therapy | Levetiracetam: Monotherapy
Number analyzed (Participants) | 32 | 6
percentage of participants | 96.9 | 100

12. Secondary Outcome: Percentage of Participants With Treatment-emergent SAEs During the Combined First and Second Period
Description: as for outcome 9
Time Frame: From Baseline (Week 0) to the End of Safety Follow-up (up to Week 295)
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Levetiracetam: Adjunctive Therapy | Levetiracetam: Monotherapy
Number analyzed (Participants) | 32 | 6
percentage of participants | 56.3 | 33.3

13. Secondary Outcome: Percentage of Participants With TEAEs Leading to Discontinuation From Study Medication During the Combined First and Second Period
Description: as for outcome 10
Time Frame: From Baseline (Week 0) to the End of Safety Follow-up (up to Week 295)
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Levetiracetam: Adjunctive Therapy | Levetiracetam: Monotherapy
Number analyzed (Participants) | 32 | 6
percentage of participants | 9.4 | 16.7

ADVERSE EVENTS:
Time Frame: From Baseline (Week 0) to the End of Safety Follow-up (up to Week 295)
Description: TEAEs were defined as those events that started on or after the date (and time) of first dose of study medication, or adverse events whose intensity worsened on or after the date (and time) of first dose of study medication. TEAEs were analyzed and reported for SS_A and SS_M.
Arm/Group | Levetiracetam: Adjunctive Therapy | Levetiracetam: Monotherapy
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/6
Serious Adverse Events (participants affected / at risk) | 18/32 | 2/6
Other Adverse Events (participants affected / at risk) | 28/32 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam: Adjunctive Therapy (N=32) | Levetiracetam: Monotherapy (N=6)
Cryptorchism (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 3 (3) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Respiratory syncytial virus bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 2 (2) | 0 (0)
Bronchitis viral (Infections and infestations) | 1 (2) | 0 (0)
Coronavirus infection (Infections and infestations) | 1 (2) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Post procedural fistula (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 3 (7) | 0 (0)
Infantile spasms (Nervous system disorders) | 3 (3) | 0 (0)
Epilepsy (Nervous system disorders) | 2 (2) | 1 (1)
Seizure cluster (Nervous system disorders) | 2 (2) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Selective eating disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epilepsy surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam: Adjunctive Therapy (N=32) | Levetiracetam: Monotherapy (N=6)
Conjunctivitis allergic (Eye disorders) | 3 (4) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 8 (10) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (10) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Dental caries (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 12 (51) | 2 (3)
Food allergy (Immune system disorders) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 17 (108) | 5 (21)
Gastroenteritis (Infections and infestations) | 7 (11) | 2 (4)
Conjunctivitis (Infections and infestations) | 6 (16) | 0 (0)
Influenza (Infections and infestations) | 5 (6) | 1 (1)
Exanthema subitum (Infections and infestations) | 5 (5) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 4 (5) | 1 (1)
Otitis media (Infections and infestations) | 3 (5) | 0 (0)
COVID-19 (Infections and infestations) | 3 (3) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 3 (3) | 3 (3)
Hordeolum (Infections and infestations) | 2 (4) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 0 (0)
Coronavirus infection (Infections and infestations) | 2 (2) | 0 (0)
Molluscum contagiosum (Infections and infestations) | 2 (2) | 1 (1)
Impetigo (Infections and infestations) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Oral contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Glucose urine present (Investigations) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 6 (7) | 0 (0)
Agitation (Psychiatric disorders) | 2 (2) | 1 (1)
Irritability (Psychiatric disorders) | 2 (2) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Balanoposthitis (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 3 (8) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (7) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Eczema (Skin and subcutaneous tissue disorders) | 9 (16) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 4 (9) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Urticaria thermal (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/64/NCT03340064/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-03): https://cdn.clinicaltrials.gov/large-docs/64/NCT03340064/SAP_001.pdf